CLINICAL TRIAL: NCT04834947
Title: Hemodynamic Effect of Prone Positioning in Non-intubated Patient With COVID 19 Pneumonia: a Monocentric Prospective Cohort Study
Brief Title: Hemodynamic Effect of Prone Position in Non-intubated Patient With COVID 19
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL21_0063
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Pneumonia, Viral
Keywords: COVID 19; prone position; hemodynamic effect; spontaneous ventilation
MeSH Terms: conditions — COVID-19; Pneumonia, Viral | interventions — Prone Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Prone position in non-intubated COVID19 , before and after.: Patients with non-intubated COVID19 pneumoniae for whom the clinician has decided to try prone positioning to increase the PaO2 in a context of hypoxemia with O2 requirement.
  Interventions: Procedure: prone position

INTERVENTIONS:
Procedure: prone position — Choice of prone positioning a patient is at the discretion of the anesthesia physician.

SUMMARY:
Prone position in non-intubated patient has shown some respiratory physiological benefits. Prone positioning in patient intubated with ARDS has shown hemodynamic benefits. We aim to compare hemodynamic assessment before and after prone positioning in non-intubated patient with COVID 19 pneumonia. The study hypothesis is that prone positioning in non-intubated patient improve right ventricular preload, reduce afterload and increase Cardiac index compared to supine position.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* COVID 19 pneumonias with Hypoxemia
* for whom prone positioning has been decided by the attending physician.

Exclusion Criteria:

* Mechanical ventilation
* ECLS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for cadiac surgery wih cardiopulmonary bypass
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-15 (Estimated); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Hemodynamic effect | Cardiac index will be recorded before, just after prone position and after return to supine position.
  Cardiac index

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Anesthésie-Réanimation, Hôpital Louis Pradel,, Bron, France